CLINICAL TRIAL: NCT04690374
Title: Registry for Patients With Desmoplastic Small Round Cell Tumor
Brief Title: Registry to Collect Health Information About Desmoplastic Small Round Cell Tumor
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20-551
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Desmoplastic Small Round Cell Tumor
Keywords: Patient registry; 20-551
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Desmoplastic small round cell tumor (DSRCT): Collect historical/longitudinal clinical, radiographic and molecular features of DSRCT patients as documented in medical records to improve knowledge about DSRCT

SUMMARY:
This study is a patient registry of people with Desmoplastic Small Round Cell Tumor (DSRCT). A patient registry is a collection of health information about a group of people, and it is usually focused on a specific diagnosis or disease.

The purpose of this registry is to create a database- a collection of information-or better understanding DSRCT. Researchers will use the information from this database to learn more about DSRCT and for current and future research on DSRCT.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of desmoplastic small round cell tumor
* Participants may be of any age as long as the appropriate consent and assent may be obtained
* Willing to provide historical and longitudinal clinical data

Exclusion Criteria:

* Participant unwilling to provide consent or share historical and longitudinal clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is a registry protocol for patients with DSRCT.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Registry to Collect Health Information About Desmoplastic Small Round Cell Tumor | 7 years
  The aim of this study is the collection of data.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm